CLINICAL TRIAL: NCT02933190
Title: Fertility After Transvaginal Surgery or Uterine Artery Embolization Combined With Uterine Curettage in Patients With Cesarean Scar Pregnancy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: ShanghaiFMIH-CSP
Record Dates: First submitted 2016-08-09; First posted 2016-10-14 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-08

CONDITIONS: Magnetic Resonance Imaging; Ovarian Function; Menstruation
MeSH Terms: interventions — Dilatation and Curettage

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (1):
- CSP；transvaginal surgery；UAE and D&C (Other): Cesarean scar pregnancy (CSP) refers to the implantation of a gestational sac with the myometrium at the site of a previous cesarean scar
  Interventions: Procedure: transvaginal surgery；UAE and D&C

INTERVENTIONS:
Procedure: transvaginal surgery；UAE and D&C — For cesarean scar pregnancy treatment

SUMMARY:
To investigate the fertility in patients after treatment by transvaginal surgery or uterine artery embolization combined with uterine curettage

ELIGIBILITY:
Inclusion Criteria:

* increased levels of serum β-hCG and ultrasonography findings. The criteria for diagnosis by ultrasonography was the presence of the following: (1) an empty uterine cavity and endocervical canal; (2) detection of the placenta and/or a gestational sac embedded in the hysterectomy scar; (3) the presence of the gestation sac with or without a fetal pole and with or without fetal cardiac activity (depending on the gestational age) in the anterior part of the uterine isthmus; and (4) a thin (1-3 mm) or absent myometrial layer between the gestational sac and the bladder(24). All patients had taken Magnetic Resonance Imaging (MRI) to clarify the diagnosis . Pregnancy tissues were identified by histopathology examinations of the surgical tissues.

Exclusion Criteria:

* All enrolled patients had no contraindications for transvaginal surgery or UAE, including renal failure, active pelvic infection, clotting disorders, or known allergy to the contrast material.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-08 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Duration of menstruation by questionnaire (days) | six months after treatment
Endocrine level by blood examination (FSH in IU/L) | six months after treatment
Volume of menstruation by questionnaire (in pictorial blood loss score) | six months after treatment

SECONDARY OUTCOMES:
The length of the CSD by MRI (millimeter) | six months after treatment
The width of the CSD by MRI (millimeter) | six months after treatment
The depth of the CSD by MRI (millimeter) | six months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Xipeng Wang, Study Chair — Department of Gynecology, Shanghai First Maternity and Infant Hospital, affiliated to Tongji University
Locations (1):
- Department of Gynecology, Shanghai First Maternity and Infant Hospital, affiliated to Tongji University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided